CLINICAL TRIAL: NCT02784665
Title: Randomized Controlled Clinical Trial to Evaluate the Effects of 577nm Micropulse Laser vs Traditional Laser Therapy on Acute Central Serous Chorioretinopathy
Brief Title: Treatment Trial for Acute Central Serous Chorioretinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jin Chen-jin (Other)
Responsible Party: Sponsor-Investigator, Jin Chen-jin, Dr, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 577MPTAC
Record Dates: First submitted 2016-05-23; First posted 2016-05-27 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Acute Central Serous Chorioretinopathy
Keywords: CSC; Micropulse Laser; Traditional Laser

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 577-MPL (Experimental): 577nm micropulse laser(577-MPL) will be performed of the areas identified on hyperfluorescent "hot spots" on the mid-phase (3 minutes) fluorescein.Multiple laser spots will be applied, covering the leakage area.
  Interventions: Device: 577-MPL
- 577-TL (Active Comparator): 577nm Traditional laser(577-TL) will be performed of the areas identified on hyperfluorescent "hot spots" on the mid-phase (3 minutes) fluorescein.Traditional laser spots will be applied, covering the leakage area.
  Interventions: Device: 577-TL

INTERVENTIONS:
Device: 577-MPL — All treatments were provided by a single practitioner with the 577-nm yellow laser system(Supra 577nm affected area in micropulse model.The power titration was started at 700 milliwatt(mW) and then gradually increased until a just visible burn was seen. When this threshold was reached, the power was reduced by 50%, using a 100-μm spot diameter and a 200-ms duration with 5 % duty cycle LaserSystem) in 577-MPL arm. The individual power for the patient was titrated at a normal area of near the
  Arms: 577-MPL
Device: 577-TL — All treatments were provided by a single practitioner with the 577-nm yellow laser system(Supra 577nm LaserSystem) in 577-TL arm.
  100 microns light spot size, 0.05 seconds duration, 80 ~ 200 milliwatts of power
  Arms: 577-TL

SUMMARY:
Central serous chorioretinopathy (CSC) is a relatively frequent eye disease in younger patients. It is characterized by serous detachment of the neurosensory retina with or without serous detachment of the retinal pigment epithelium (RPE), which can cause vision drop, image distortion, loss of color and contrast vision. Although nonfoveal focal leakage can be treated with traditional laser photocoagulation, but it has the side effects of causing RPE atrophy, scotoma, or secondary CNV. Photodynamic therapy (PDT) is another effective treatment but it's more than most families can afford to pay because of the high cost, what's more, it is accompanied with side-effects, such as choroidal ischemia, retinal pigmental epithelium (RPE) atrophy and RPE rip.

To date there is no international consensus on the optimal treatment of CSC Many retrospective studies suggest that micropulse laser (MPL) therapy may also be effective without obvious complications in this disease.

The purpose of this study is to evaluate the effect of micropulse laser (MPL) on acute central serous chorioretinopathy compared with the traditional laser coagulation.

DETAILED DESCRIPTION:
The study is a prospective randomized controlled trial about 577nm micropulse laser versus traditional laser coagulation therapy on acute central serous chorioretinopathy. The primary outcome measures is the proportion of eyes with complete absorption of subretinal fluid 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. onset for the first time, as an episode duration of less than 6 months
2. patient was between 18 and 55 years of age
3. the presence of subretinal fluid(SRF) involving the macula and detected by use of optical coherence tomography (OCT)
4. active fluorescein leakage during fluorescein angiography (FA)
5. best corrected visual acuity (BCVA) more than 0.1, and less than 1.0

Exclusion Criteria:

1. previous PDT, focal photocoagulation, intravitreal injections of anti-vascular endothelial growth factor, or ocular surgery
2. other macular abnormalities such as choroidal neovascularization(CNV) or polypoidal choroidal vasculopathy(PCV)
3. retinal atrophy
4. pregnancy
5. inability to obtain photographs or to perform FA
6. use of steroid systemically or topically in the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
the proportion of eyes with complete absorption of subretinal fluid (SRF) | 3 month
  The primary outcome measure is the OCT-based improvement rate (defined as the proportion of eyes with complete absorption of subretinal fluid on OCT images)

SECONDARY OUTCOMES:
Change of Best Corrected Visual Acuity (BCVA) | 1months,3 months and 6 months
Change of fundus autofluorescence | 1months,3 months and 6 months
  Fundus autofluorescence will be evaluated for different patterns (normal, increased, and decreased) before and after treatment
Change in 10° retinal sensitivity | baseline,1months,3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided